CLINICAL TRIAL: NCT00604981
Title: Adapting Multisystemic Therapy to Improve Food Choices and Health Outcomes in Obese African American Youth
Brief Title: Multisystemic Therapy (MST) for Obesity in African American Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sylvie Naar-King, Ph.D., Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7-05-HFC-24
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Multisystemic Therapy (MST)
  Interventions: Behavioral: Multisystemic Therapy (MST)
- 2 (Active Comparator): Shapedown
  Interventions: Behavioral: Shapedown

INTERVENTIONS:
Behavioral: Multisystemic Therapy (MST) — MST is an intensive, family centered, community based treatment originally designed for use with adolescents presenting with serious mental health problems. In this study, MST interventions are aimed at increasing adolescent and family adherence to dietary and exercise recommendations and targeting barriers within the family system, and the broader community systems within which the family is embedded (peers, schools, health care). Decreasing caloric consumption consistent with recommended intake targets, increasing daily exercise and decreasing sedentary activity, are treatment focuses depending on whether the adolescent has difficulty with this aspect of weight management or not.
  Arms: 1
Behavioral: Shapedown — Shapedown, is a clinic-based, adolescent weight loss intervention. Shapedown utilizes psycho educational, behavior, and family therapy techniques in a 10-week group intervention. In order to match MST's length of intervention (6 months), three follow-up sessions are added at monthly intervals.
  Arms: 2

SUMMARY:
Despite the dramatic increase in obesity and Type II Diabetes in adolescents, documented effective treatments for obesity and the consequential prevention of Type II Diabetes are scarce. Modification of food and activity choices is the foundation of obesity treatment; however, adolescents may find it difficult to follow recommended diet and exercise programs. This study uses a home-based treatment, Multisystemic Therapy (MST), to target change within the individual, family and environmental contexts. Participants are 49 obese (BMI>95th percentile) African American adolescents (ages 12-17). 24 were randomized to receive the MST intervention and 25 were placed in Shapedown, a family group program. Families were recruited from the only university-affiliated medical center in Detroit, Michigan. Michigan's youth have higher rates of obesity, overweight, hypertension, and elevated cholesterol compared to the national average, and Detroit has the highest percentage of African Americans of any major city in the US. Families complete measurements at the start of the treatment, at the end of the treatment and one year after enrollment. We expect to find that youth in the MST group will show more weight loss and greater improvements in diet (e.g., caloric intake and exercise behaviors than will youth in Shapedown. These changes in food choices, activity levels, and weight are expected to remain after the end of treatment. This intervention is intended to provide immediate assistance to a vulnerable population disproportionately affected by obesity and its long-term health complications.

DETAILED DESCRIPTION:
Despite the increase in pediatric obesity, controlled intervention trials among adolescents are rare and fail to address vital socio-ecological factors, particularly in minority youth. Modification of food and activity choices is the foundation of obesity treatment; however, adherence to these recommendations is a major barrier. We have adapted the home-based Multisystemic Therapy (MST) to successfully improve outcomes in urban adolescents with diabetes. The objective of the present study is to adapt MST to improve adherence to recommended food and activity choices and reduce BMI in obese (BMI>95th percentile) African American adolescents (ages 12-17). Additional aims are to determine if MST changes the individual, family, and environmental variables related to poor food choices (e.g., parental monitoring). Families are recruited from the only university-affiliated medical center in Detroit, Michigan. Michigan's youth have higher rates of obesity, overweight, hypertension, and elevated cholesterol compared to the national average. Detroit has the highest percentage of African Americans of any major city in the US. The design is a randomized controlled trial with 49 obese African American adolescents, 24 of whom receive MST and 25 of whom receive Shapedown, a family-based behavioral group intervention. Families complete a baseline data collection, a 7-month post-test coinciding with treatment completion, and a 12-month post-test. The primary aim of this project is Despite the increase in pediatric obesity, controlled intervention trials among adolescents are rare and fail to address vital socio-ecological factors, particularly in minority youth. Modification of food and activity choices is the foundation of obesity treatment; however, adherence to these recommendations is a major barrier. We have adapted the home-based Multisystemic Therapy (MST) to successfully improve outcomes in urban adolescents with diabetes. The objective of the present study is to adapt MST to improve adherence to recommended food and activity choices and reduce BMI in obese (BMI>95th percentile) African American adolescents (ages 12-16). Additional aims are to determine if MST changes the individual, family, and environmental variables related to poor food choices. Families will be recruited from the only university-affiliated medical center in Detroit, Michigan. Michigan's youth have higher rates of obesity, overweight, hypertension, and elevated cholesterol compared to the national average. Detroit has the highest percentage of African Americans of any major city in the US. The design is a randomized controlled trial with 49 obese African American adolescents, 24 of whom receive MST and 25 of whom receive a family-based behavioral group intervention. Families complete a baseline data collection, a 7-month post-test coinciding with treatment completion, and a 12-month post-test. If successful, this intervention will provide immediate assistance to a vulnerable population disproportionately affected by obesity and its long-term health complications. The project will also provide the foundation for a larger clinical trial as well as future interdisciplinary studies combining behavioral and medical interventions. If successful, this intervention will provide immediate assistance to a vulnerable population disproportionately affected by obesity and its long-term health complications. The project will also provide the foundation for a larger clinical trial as well as future interdisciplinary studies combining behavioral and medical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Primary obesity as indicated by a BMI percentile >=95th based on current height and weight using age and gender norms from the Centers for Disease Control and Prevention
* Self-identified as African American
* Between the ages of 12 years, 0 months and 17 years, 11 months and
* Residing in a home environment with a caregiver who was willing to participate in treatment.

Exclusion Criteria:

* Pregnancy
* Moderate or severe mental retardation or psychosis; AND
* Medical co morbidities that required treatment, including diabetes and hypertension.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
weight (lbs, BMI) | baseline, 7 months post treatment, 12 months post treatment

SECONDARY OUTCOMES:
food choices | baseline, 7 months (post treatment), 12 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Pediatric Prevention Research Center, Detroit, Michigan, United States